CLINICAL TRIAL: NCT05574192
Title: Building Supportive Social Networks to Advance the Mental Health of Women Affected by Violence in Vancouver's Downtown East Side
Brief Title: The Social Engagement Project: Addressing Isolation with Women Affected by Violence
Acronym: SEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Inner-City Women's Initiatives Society (Unknown); Vancouver Foundation (Other)
Responsible Party: Principal Investigator, Victoria Bungay, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H22-02504
Record Dates: First submitted 2022-09-29; First posted 2022-10-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Loneliness; Social Support; Social Isolation
Keywords: peer-led intervention; mixed-method; community-based; vulnerable women; supportive social networks; gender-based violence
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Mixed-method participatory action research design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Social Engagement Intervention (Other): The social engagement intervention includes in-person visits by peer-workers to undertake accompanied social activities with enrolled participants. Each visit will last one hour, occur two times per month over a 12 month period. Activity categories will be self-selected by participants based on physical abilities and interests. Categories include: a) arts based activity; b) physical activity.
  Interventions: Behavioral: Social Engagement Intervention

INTERVENTIONS:
Behavioral: Social Engagement Intervention — The intervention includes social visiting with women affected by violence. Social visiting is carried out by trained peer-workers. Peers are women who share life histories with the target study population. Peer-workers will establish a visiting schedule (day/time) and provide a detailed list of activities in two categories:
  1. arts-based activities.
  2. physical activities.
  The peer will meet with the participant at the scheduled place and times to accompany the participant and engage in the activities with the participant.
  Participation in scheduled social activities that target the interest and ability of women affected by violence is considered to improve social connectedness by increasing the quality and quantity of a woman's social interactions with a supportive, trained person who shares life experiences. Shared, consistent and reliable social activities also are hypothesized to reduce loneliness by contributing to a sense of belonging and sense of being cared for.

SUMMARY:
The goal of this study is to test a pilot intervention aimed at improving social connectedness among women affected by gender-based violence in a resource-restricted, urban context. The intervention will specifically address barriers to building and sustaining supportive social networks to reduce women's risks for worsening mental health associated with isolation, with a focus on barriers stemming from gender-based violence and poverty. The main question it aims to answer are:

* How acceptable is the intervention to women affected by gender-based violence including the benefits, burdens and appropriateness in the context of their everyday lives?
* How feasible is the intervention and study protocol?
* What are the effects of a peer-led social engagement intervention to develop and sustain supportive social networks and reduce isolation among women affected by gender-based violence?

Participants will engage in social activities with trained peer workers over a one-year period.

DETAILED DESCRIPTION:
This study is designed to assess feasibility, acceptability, and preliminary effects of a behavioral intervention aimed at improving social connectedness among women affected by gender-based violence in a resource-restricted, urban context through a pilot intervention using a case study design informed by principles of community-based participator action research. The intervention is a peer-led social visiting program delivered over a 12 month period. Primary outcomes include feasibility (recruitment, retention) and acceptability (timing and frequency of social activities, perceived satisfaction). The investigators will also determine whether the intervention shows the potential to increase social connectedness over a 12-month period.

Population Adult women living in a dense, urban context where poverty, precarious housing and problematic substance use are evident who are at risk of or living with gender-based violence.

Objectives The goal of this work is to test the feasibility, acceptability and preliminary effects of the intervention on social connectedness among women affected by gender-based violence.

The primary objectives are to assess:

1. Acceptability of the intervention to participants, peer-support workers, and staff.
2. Feasibility of delivering the intervention within a resource-restricted setting where participants are experiencing severe poverty and other forms of disadvantage such as mental health challenges, complex physical health concerns, and violence.

The secondary objectives are to measure the intervention's effect on social connectedness and its related elements (loneliness, socializing, social support, and sense of belonging) at 12-months.

Endpoints

The endpoints for the primary objectives:

1. Quantitative and qualitative reports of intervention acceptability among participants; quantitative and qualitative reports of acceptability among peer-support workers (intervention providers); qualitative reports of acceptability among staff managing the peer-support workers.
2. Measures of feasibility include recruitment, retention, intervention participation, financial cost, and fidelity of intervention delivery.

The endpoints for the secondary objective are specific to the elements of social connectedness and include qualitative and quantitative reports of perceived sense of loneliness, social support, and sense of belonging; quantitative reports of attendance at social activities; quantitative reports of social networks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Self-identify as a woman (trans-inclusive);
3. Able to verbally communicate in English;
4. Have a consistent place to live that is not a temporary shelter;
5. Have lived in the same place for at least one month;
6. Live and/or spend significant time for work and/or health and social services in the study catchment area
7. Able and willing to provide adequate contact information Age 18 or over
8. Willing and able to provide consent

Exclusion Criteria:

1. planning to travel away from the study catchment area for a time period that would interfere with study participation;
2. is experiencing a condition that, in the opinion of the site PI, would preclude informed consent or make study participation unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants self-identify as a woman.
Enrollment: 42 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention - qualitative data from participants | 2 months
  Acceptability measures include qualitative reports of intervention acceptability among participants. These will include in-depth interviews to explore goals and rationale for enrolling in the intervention as well as expectations and perspectives about initial social engagement activities
Acceptability of the intervention - qualitative data from participants | 12 months
  Acceptability measures include qualitative reports of the intervention acceptability among participants. Upon intervention completion, in-depth qualitative interviews covering topics such as satisfaction with the content, length, and delivery of the intervention as well as reported impact on participants' life
Acceptability of the intervention - quantitative data from participants [survey tool] | 6 months
  Satisfaction with intervention content,delivery, length, using a survey tool and measured on a likert scale response 1 to 5 with higher indicating higher satisfaction and as open ended response options
Acceptability of the intervention - quantitative data from participants [survey tool] | 12 months
  Satisfaction with intervention content,delivery, length, using a survey tool and measured on a likert scale response 1 to 5 with higher indicating higher satisfaction an as open ended responses
Acceptability of intervention - qualitative data from peer workers | 3 months
  Acceptability measures include qualitative reports of the intervention acceptability among peer support workers. These will include in-depth qualitative interviews about the delivery and length of the intervention.
Acceptability of intervention - qualitative data from peer workers | 12 months
  Acceptability measures include qualitative reports of the intervention acceptability among peer support workers. These will include in-depth qualitative interviews
Acceptability of the intervention - qualitative data from staff | 12 months
  Acceptability measures include qualitative reports of the intervention acceptability among peer support workers. These will include in-depth qualitative interviews about the implementation process, the content, timing and delivery of the intervention.
Feasibility of the intervention - Retention - forms | 12 months
  proportion of participants who complete initial enrollment, retention is >75% at 12 months
Feasibility of the intervention - process fidelity - forms | throughout the study; 12 months
  observations of intervention delivery capturing activities administered;
Feasibility of the intervention - financial cost - forms | 12 months
  calculated total cost for intervention activities; total cost calculated using cash amounts for salaries of providers and intervention activities. Time frame. 12 months
Feasibility of the Intervention - qualitative data from staff | 12 months
  Feasibility includes qualitative reports of the strengths and challenges experienced implementing a behavioural intervention in a community setting. In-depth interviews with staff will explore the specific experiences of implementing peer-led initiatives with women affected by violence who are living in extreme poverty and experience numerous physical and mental health challenges.

SECONDARY OUTCOMES:
Social Connectedness - survey tool | 2 weeks
  Self-report experiences of social connectedness in the past 3 months using questions about frequency of social activities with others (total number experienced), sense of belonging in community (likert scale response with higher being greater sense of belonging), and perceived social support with questions about the quality of relationships with others (likert scale with lower score indicating higher quality).
Social Connectedness - survey tool | 6 months
  Self-report experiences of social connectedness in the past 3 months using questions about frequency of social activities with others in the past 3 months (total number experienced), sense of belonging in community (likert scale response with higher being greater sense of belonging), and perceived social support with questions on questions about the quality of relationships with others (likert scale with lower score indicating higher quality).
Social Connectedness - survey tool | 12 months
  Self-report experiences of social connectedness in the past 3 months using questions about frequency of social activities with others in the past 3 months (total number experienced), sense of belonging in community (likert scale response with higher being greater sense of belonging), and perceived social support with questions on questions about the quality of relationships with others (likert scale with lower score indicating higher quality).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bungay, Principal Investigator — The University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No